CLINICAL TRIAL: NCT01650285
Title: Cabazitaxel and Radiation For Patients With Pathologically Determined Stage 3 Prostate Cancer and/or Patients With PSA Elevation (>0.1- < 2.0 ng/mL) Following Radical Prostatectomy
Brief Title: Cabazitaxel and Radiation For Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment and lost funding
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 246
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel and radiation (Experimental): Radiation therapy (RT) will be delivered to 64.8 Gy, using IMRT treatment Cabazitaxel will be administered IV every 21 days for 3 doses at the assigned dose level.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Dose Level Day 1, 22, 43
  1. 5.0 mg/m2
  2. 10.0 mg/m2
  3. 15.0 mg/m2
  4. 20.0 mg/m2
  Other Names: Jevtana

SUMMARY:
There is a high relapse rate for patients who have undergone prostatectomy and have pathologic extracapsular prostate extension, positive surgical margins or seminal vesicle involvement (pathologic stage 3 disease). While adjuvant radiation improves progression-free and overall survival, approximately half of these patients will develop recurrence. Similarly, radiation therapy has become the standard salvage therapy for patients with rising PSA >0.1 - < 2.0 ng/mL. In common solid tumors such as NSCLC, head and neck cancer and upper gastrointestinal cancers, the addition of chemotherapy to radiation improves survival. It is hypothesized that the addition of radiosensitizing chemotherapy to standard adjuvant radiation will improve survival in patients with stage 3 prostate cancer after prostatectomy and patients with rising PSA < 2.0 ng.mL without detectable disease. Taxanes are powerful radiation enhancers since they synchronize tumor cells in G2/M the most radiosensitive phase of the cell cycle.17,18 Cabazitaxel is the most active taxane in the treatment of prostate cancer. Therefore, we propose a phase I study establishing the optimal dose of cabazitaxel with adjuvant radiation for stage 3 prostate cancer after prostatectomy (PSA undetectable - < 2.0 ng/mL). and for patients with persistent or rising PSA post prostatectomy (PSA >0.1 - < 2.0 ng/mL).

ELIGIBILITY:
Conditions for Patient Eligibility

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Radical prostatectomy for adenocarcinoma of the prostate with at least one of the following:

  * Extracapsular tumor extension,
  * Positive surgical margins,
  * Seminal vesicle invasion
  * Regional lymph node positive (N1)
  * Post-prostatectomy PSA of > 0.1 - < 2.0 ng/mL at least 6 weeks after prostatectomy and within 30 days of registration in a patient with T2 or T3 disease at prostatectomy.
* No distant metastases.
* No prior pelvic or prostate radiation or chemotherapy for prostate cancer.
* ECOG performance status 0-1.
* Age>18.
* Required entry laboratory parameters within 14 days of study entry: Granulocytes ≥ 1500 cells/mm3; platelet count ≥100,000 cells/mm3, Creatinine ≤ 1.5X upper limit of normal (if creatinine clearance 1.0-1.5x ULN, creatinine clearance will be calculated according to Chronic Kidney Disease Epidemiology Group formula and patients with creatinine clearance < 60 ml/min should be excluded),19 .Hgb > 9.0 g/dl, total bilirubin ≤ 1x ULN, and AST or ALT ≤ 2.5 x ULN.
* Life expectancy of at least 1 year.
* Must not have uncontrolled severe, intercurrent illness.
* No concurrent anticancer therapy.
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Signed study-specific consent form prior to study entry.
* Conditions for Patient Ineligibility

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Evidence of distant metastases (M1). Equivocal bone scans are allowed if plain films are negative for metastasis.
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the oral cavity or bladder are permissible).
* History of severe hypersensitivity (> grade 3) reaction to Cabazitaxel or other drugs formulated with polysorbate 80.
* History of severe hypersensitivity (> grade 3) to docetaxel.
* Any uncontrolled severe, intercurrent illness (including uncontrolled diabetes)
* At least 4 weeks since any major surgery.
* Patients on concurrent anticancer therapy.
* PSA > 2ng/ml
* Concurrent or planned treatment with strong inhibitors or inducers of cytochrome p450 3A4/5 (a one-week wash out period is necessary for patients who are already on these treatments (see appendix H and I)
* Androgen deprivation therapy started prior to prostatectomy for > 6 months duration;
* Neoadjuvant chemotherapy prior to prostatectomy;
* Prior cryosurgery or brachytherapy of the prostate; prostatectomy should be the primary treatment and not a salvage procedure;
* Prior pelvic radiotherapy;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — Brown University; anthony mega, md, Principal Investigator — Lifespan
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabazitaxel and Radiation: Radiation therapy (RT) will be delivered to 64.8 Gy, using IMRT treatment Cabazitaxel will be administered IV every 21 days for 3 doses at the assigned dose level.
  Cabazitaxel: Dose Level Day 1, 22, 43
  1. 5.0 mg/m2
  2. 10.0 mg/m2
  3. 15.0 mg/m2
  4. 20.0 mg/m2
Period: Overall Study
Arm/Group | Cabazitaxel and Radiation
Started | 5
Completed | 4
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cabazitaxel and Radiation
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 61 [56 to 64]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Cabazitaxel With Concurrent Adjuvant Radiation
Description: The MTD was not determined secondary to the study closing early. That being said the numbers provided below show that 4 patients were treated on study to aide in the investigation of the MTD. Only 1 dose was fully evaluated which was 5mg/m2
Time Frame: 2 mos
Population: while 5 participants were enrolled only 4 completed treatment as patients # 5 only received part of day 1 therapy secondary to an AE and therefore is not included in the assessment.
Measure: Number; unit: mg/m2
Arm/Group | Cabazitaxel and Radiation
Number analyzed (Participants) | 4
mg/m2 | NA — only the 5mg/m2 dose was evaluated due to the study closing early and MTD was not determined)

2. Secondary Outcome: Number of Participants Experiencing a Toxicity Associated With Cabazitaxel and Adjuvant Radiation Following Prostatectomy for Patients With Stage 3 Prostate Cancer and for Patients With a PSA Elevation Post-Prostatectomy.
Description: Assess toxicity using CTCAE version 4.0. Number of patients who experienced a toxicity on the study. Not all toxicities are related to study treatment. Of note, there were no serious adverse events on this trial.
Time Frame: During study treatment (approximately 8 weeks) through 30 days post treatment, approximately 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabazitaxel and Radiation
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: From time of informed consent to approximately 30 days post last dose of drug- approximately 3 months.
Arm/Group | Cabazitaxel and Radiation
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel and Radiation (N=5)
anemia (Investigations) | 2 (2)
anorexia/decreased appetite (Investigations) | 2 (2)
constipation (Investigations) | 1 (1)
diarrhea (Investigations) | 3 (3)
dizziness (Investigations) | 1 (1)
fatigue (Investigations) | 5 (5)
flatulence (Investigations) | 1 (1)
GI Hemorrhage (Investigations) | 1 (1)
glucose (Investigations) | 2 (2)
hemmorhoids (Investigations) | 1 (1)
Hot flashes (Investigations) | 2 (2)
Hypersensitivity rxn (Investigations) | 1 (1)
Potassium (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
myalgia/ malaise (Investigations) | 1 (1)
nausea (Investigations) | 2 (2)
Pain- leg (Investigations) | 1 (1)
pain-abdominal (Investigations) | 1 (1)
urinary frequency (Investigations) | 2 (2)
WBC (Investigations) | 1 (1)
Aches (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No